CLINICAL TRIAL: NCT07120828
Title: The Role of CYP8B1 Polymorphisms in Modulating the Biochemical Pathways Affected by SGLT2 Inhibitors in T2DM and Obesity
Acronym: CYP8B1-SGLT2-T
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erbil Polytechnic University (Other)
Collaborators: Kurdistan Higher Council of Medical Specialties (Other)
Responsible Party: Principal Investigator, Ahmed Abdulrazzaq Bapir, PhD Student (under supervision of Prof. goran othman ), Kurdistan Higher Council of Medical Specialties
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPU-CYP8B1-SGLT2-T2DM-2025-01; No: 2348524, February 21, 2025 (Other: Salahaddin University-Erbil)
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Obese Diabetics; Obese Patients (BMI ≥ 30 kg/m²)
Keywords: CYP8B1; Obese diabetics; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Empagliflozin Group (Experimental): Participants in this group will receive empagliflozin 10 mg orally once daily for a duration of 6 months. The intervention aims to evaluate the effect of empagliflozin on weight reduction, metabolic parameters, and biochemical outcomes in newly diagnosed obese T2DM patients, with a focus on the influence of CYP8B1 polymorphisms on treatment response.
  Interventions: Drug: Empagliflozin (oral)
- Dapagliflozin Group (Experimental): Participants in this group will receive dapagliflozin 10 mg orally once daily for a duration of 6 months. This arm is designed to assess the clinical and biochemical effects of dapagliflozin, particularly regarding changes in adipokines, lipid profile, insulin sensitivity, and the impact of CYP8B1 genetic variations.
  Interventions: Drug: Dapagliflozin (DAPA)
- Control Group (Active Comparator): Participants in this group will receive standard care, including dietary and lifestyle modifications and metformin therapy if clinically indicated, according to ADA guidelines. This arm will serve as a comparator to evaluate the relative efficacy of SGLT2 inhibitors and the role of CYP8B1 polymorphisms in treatment outcomes.
  Interventions: Drug: Metfomin

INTERVENTIONS:
Drug: Empagliflozin (oral) — Empagliflozin 10 mg oral tablet administered once daily for 6 months.
  Arms: Empagliflozin Group
Drug: Dapagliflozin (DAPA) — Dapagliflozin 10 mg oral tablet administered once daily for 6 months
  Arms: Dapagliflozin Group
Drug: Metfomin — metformin 500-1000 mg/day administered as part of standard care, based on clinical indication.
  Arms: Control Group

SUMMARY:
This study explores the long-term effects of dapagliflozin and empagliflozin on CYP8B1 gene expression and a range of metabolic, oxidative, and inflammatory biomarkers in obese patients with Type 2 Diabetes Mellitus (T2DM). Over a 6-month period, participants are assigned to three treatment arms: metformin (control), dapagliflozin, and empagliflozin. The study aims to determine how these medications influence bile acid metabolism, oxidative stress, leptin, GLP-1, IL-10, and IFN-γ, providing insight into the broader metabolic benefits of SGLT2 inhibitors

DETAILED DESCRIPTION:
Detailed Description Type 2 Diabetes Mellitus (T2DM) and obesity are major global health burdens with shared pathophysiological mechanisms, including insulin resistance, chronic inflammation, and altered lipid metabolism. SGLT2 inhibitors, such as empagliflozin and dapagliflozin, have emerged as effective glucose-lowering agents that also offer additional benefits, including weight reduction, cardiovascular protection, and renal function preservation.

Despite these advantages, the therapeutic response to SGLT2 inhibitors is variable, often influenced by individual genetic differences. A key genetic determinant is CYP8B1 (cytochrome P450 family 8 subfamily B member 1), a gene encoding sterol 12-alpha-hydroxylase, which regulates bile acid synthesis and lipid metabolism. Polymorphisms in CYP8B1 may impact drug metabolism and alter bile acid-mediated metabolic regulation, potentially affecting both the efficacy and safety profile of SGLT2 inhibitors.

This clinical trial aims to investigate the role of CYP8B1 genetic variations in modifying the clinical and biochemical responses to empagliflozin and dapagliflozin therapy among obese patients recently diagnosed with T2DM.

Participants will be randomized into three groups:

* Group 1: Empagliflozin 10 mg daily
* Group 2: Dapagliflozin 10 mg daily
* Group 3 (Control): Standard care (lifestyle modification and/or metformin)

The intervention period is 6 months, during which multiple parameters will be monitored:

1. Obesity-Related Metrics: Body weight, BMI, waist circumference, and body fat percentage.
2. Adipokines: adiponectin.
3. Lipid Profile: Total cholesterol, HDL, LDL, and triglycerides.
4. Glycemic Control: Fasting glucose, HbA1c, and C-peptide.
5. Oxidative Stress & Inflammation
6. Ketone Bodies & Free Fatty Acids: To assess shifts in metabolic fuel utilization.
7. Insulin Sensitivity: Using QUICKI and Adipo-IR indices.
8. CYP8B1 Genotyping & Expression: PCR-based genotyping and qPCR-based expression profiling to evaluate genetic and transcriptional regulation.

   The study integrates molecular genetics (Sanger sequencing and RT-PCR) with clinical biochemistry and metabolic phenotyping to provide a holistic understanding of pharmacogenomic effects.

   Expected outcomes include:

   • Determining whether CYP8B1 polymorphisms influence the degree of weight loss, lipid and glucose metabolism, and adipokine modulation.
   * Comparing the efficacy of empagliflozin vs dapagliflozin in the presence of different CYP8B1 genotypes.
   * Proposing a framework for personalized T2DM and obesity management based on genetic screening.

   Study Type Observational Clinical Trial

   ________________________________________ Study Duration Estimated Study Period: 6 months per participant

   ________________________________________ Eligibility Criteria

   Inclusion Criteria:
   * Aged ≥18 years
   * Newly diagnosed T2DM (<6 months)
   * BMI ≥30 kg/m²
   * No prior antidiabetic treatment
   * Consent to genetic testing

   Exclusion Criteria:

   • Type 1 diabetes or secondary diabetes

   • Severe renal impairment (eGFR <45 mL/min/1.73 m²)

   • Liver dysfunction or active liver disease
   * Pregnancy or lactation
   * Allergy to SGLT2 inhibitors

   Primary Outcome Measures

   • Change in body weight and BMI at 6 months
   * Genotype-specific differences in weight loss Secondary Outcome Measures
   * Changes in adipokine levels
   * Lipid profile changes
   * HbA1c and fasting blood glucose improvement
   * Differences in insulin sensitivity indices
   * Expression levels of CYP8B1 mRNA
   * Relationship between genotype and biochemical/metabolic outcomes

   Statistical Analysis Plan
   * Paired t-tests and ANOVA for within-group and between-group comparisons
   * Genotype-phenotype association using chi-square and regression models
   * ROC curve analysis for predicting treatment response
   * Cox regression for time-to-event data

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Type 2 Diabetes Mellitus (within the past 6 months).
* Body Mass Index (BMI) ≥ 30 kg/m² (classified as obese).
* No prior treatment with SGLT2 inhibitors or other antidiabetic medications.
* Willing and able to provide written informed consent.
* Able to comply with study visits, procedures, and sample collection.

Exclusion Criteria:

* History or diagnosis of Type 1 diabetes mellitus or secondary forms of diabetes.
* Estimated Glomerular Filtration Rate (eGFR) < 45 mL/min/1.73 m² (moderate to severe renal impairment).
* Active liver disease or significant hepatic dysfunction.
* Current pregnancy or breastfeeding.
* Known hypersensitivity or contraindication to SGLT2 inhibitors.
* hypertension
* Any other condition that, in the opinion of the investigator, may interfere with the patient's ability to complete the study or pose additional risk.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight (kg) from Baseline to 6 Months | Baseline and 6 months
  Body weight will be measured using a calibrated digital scale at baseline and at 6 months. The change in weight will be calculated by subtracting baseline weight from 6-month weight.
Change in Serum Total Cholesterol (mg/dL) from Baseline to 6 Months | Baseline to 6 Months
  Serum total cholesterol will be measured using standard enzymatic methods at baseline and after 6 months. The change will be calculated by subtracting baseline values from follow-up values.
Change in Malondialdehyde (MDA) Levels (µmol/L) from Baseline to 6 Months | Baseline to 6 Months
  Serum MDA will be measured using the TBARS assay to assess lipid peroxidation and oxidative stress.
CYP8B1 Gene Expression Changes | Baseline to 6 Months
  Measure CYP8B1 mRNA expression using real-time PCR to evaluate the relationship between gene expression and treatment response.

SECONDARY OUTCOMES:
Change in Adiponectin Levels | Baseline to 6 Months
  determine changes in serum adiponectin (ng/mL) levels and evaluate their correlation with treatment response and CYP8B1 genotype.
Change in HbA1c | Baseline to 6 Months
  Measure glycated hemoglobin (HbA1c, %) to evaluate the effectiveness of SGLT2 inhibitors in glycemic control in relation to CYP8B1 polymorphisms.
Change in Fasting Blood Glucose | Baseline to 6 Months
  Determine the impact of interventions on fasting glucose levels (mg/dL).
Change in C-Peptide Levels | Baseline to 6 Months
  Evaluate β-cell function by analyzing fasting C-peptide concentrations (ng/mL) pre- and post-treatment.
Change in Blood Ketone Body Levels | Baseline to 6 Months
  Quantify changes in serum ketone levels (mmol/L) to assess shifts in energy metabolism.
Change in Serum HDL Cholesterol (mg/dL) from Baseline to 6 Months | Baseline and 6 Months
  Serum HDL cholesterol will be measured using direct enzymatic assay at baseline and 6 months to evaluate changes in HDL levels.
change in Serum LDL Cholesterol (mg/dL) from Baseline to 6 Months | Baseline and 6 Months
  LDL cholesterol will be calculated using the Friedewald equation , and compared between baseline and 6-month values
Change in Serum Triglycerides (mg/dL) from Baseline to 6 Months | Baseline and 6 Months
  Serum triglyceride levels will be measured enzymatically at baseline and 6 months to assess changes.
Change in Superoxide Dismutase (SOD) Activity (U/mL) from Baseline to 6 Months | Baseline and 6 Months
  SOD enzyme activity will be measured in serum using a colorimetric assay to evaluate antioxidant defense status at baseline and 6 months.
Change in Serum Interleukin-10 (IL-10) Levels (pg/mL) from Baseline to 6 Months | Baseline to 6 Months
  IL-10 will be quantified using a high-sensitivity ELISA kit in serum samples collected at baseline and 6 months.
Change in Glutathione Peroxidase (GPx) Activity (U/mL) from Baseline to 6 Months. | Baseline to 6 Months
  GPx enzyme activity will be measured in serum using a colorimetric assay to evaluate antioxidant defense.
Change in Catalase Activity (U/mL) from Baseline to 6 Months | Baseline to 6 Months
  Catalase activity in serum will be assessed using a spectrophotometric assay to evaluate antioxidant capacity.
Change in Interferon-Gamma (IFN-γ) Levels (pg/mL) from Baseline to 6 Months | Baseline to 6 Months
  Serum IFN-γ levels will be measured using enzyme-linked immunosorbent assay (ELISA) to assess pro-inflammatory status.
Change in Nitric Oxide (NO) Levels (µmol/L) from Baseline to 6 Months | Baseline and 6 Months
  Nitric oxide concentration will be determined in serum using the Griess reaction to evaluate nitrosative stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Epu, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: No
The data collected in this study will not be shared due to institutional policies, ethical concerns, and protection of participant confidentiality.

REFERENCES:
- [Background] Scheen AJ. Sodium-glucose cotransporter type 2 inhibitors for the treatment of type 2 diabetes mellitus. Nat Rev Endocrinol. 2020 Oct;16(10):556-577. doi: 10.1038/s41574-020-0392-2. Epub 2020 Aug 27. PMID 32855502
- [Background] Malone JI, Hansen BC. Does obesity cause type 2 diabetes mellitus (T2DM)? Or is it the opposite? Pediatr Diabetes. 2019 Feb;20(1):5-9. doi: 10.1111/pedi.12787. Epub 2018 Nov 5. PMID 30311716
- [Background] Klen J, Dolzan V. Treatment Response to SGLT2 Inhibitors: From Clinical Characteristics to Genetic Variations. Int J Mol Sci. 2021 Sep 10;22(18):9800. doi: 10.3390/ijms22189800. PMID 34575958
- [Background] Hegyi P, Maleth J, Walters JR, Hofmann AF, Keely SJ. Guts and Gall: Bile Acids in Regulation of Intestinal Epithelial Function in Health and Disease. Physiol Rev. 2018 Oct 1;98(4):1983-2023. doi: 10.1152/physrev.00054.2017. PMID 30067158
- [Background] Fioretto P, Zambon A, Rossato M, Busetto L, Vettor R. SGLT2 Inhibitors and the Diabetic Kidney. Diabetes Care. 2016 Aug;39 Suppl 2:S165-71. doi: 10.2337/dcS15-3006. PMID 27440829
- [Background] Chiang JYL, Ferrell JM. Bile Acids as Metabolic Regulators and Nutrient Sensors. Annu Rev Nutr. 2019 Aug 21;39:175-200. doi: 10.1146/annurev-nutr-082018-124344. Epub 2019 Apr 24. PMID 31018107
- [Background] Chiang JY. Bile acid metabolism and signaling. Compr Physiol. 2013 Jul;3(3):1191-212. doi: 10.1002/cphy.c120023. PMID 23897684
- [Background] Sarafidis PA, Tsapas A. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1092. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981941